CLINICAL TRIAL: NCT03065075
Title: Effect of Phenazopyridine on Prolapse Surgery Voiding Trials
Acronym: EPOV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Michael Flynn, MD, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H00012082
Record Dates: First submitted 2017-02-10; First posted 2017-02-27 (Actual); Results first posted 2019-03-26 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Urinary Retention Postoperative
MeSH Terms: interventions — Phenazopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenazopyridine (Experimental): Participant is given Phenazopyridine 200mg on postoperative day 1
  Interventions: Drug: Phenazopyridine
- No Phenazopyridine (No Intervention): Participant is not given Phenazopyridine on postoperative day 1

INTERVENTIONS:
Drug: Phenazopyridine — Phenazopyridine 200 mg on morning of postoperative day 1
  Other Names: Pyridium
  Arms: Phenazopyridine

SUMMARY:
To determine if phenazopyridine reduces the rate of postoperative urinary retention after pelvic organ prolapse surgery.

DETAILED DESCRIPTION:
Several tools can be used to evaluate for ureteral patency during urogynecologic procedures. Typically, surgeons use urine dyes such as methylene blue, indigotindisulfonate sodium, or phenazopyridine, with the latter being restricted to oral administration. However in June 2014, the two U.S. manufacturers of indigotindisulfonate sodium stopped producing the medication and there is no prospect that it will be returning soon. Phenazopyridine is an over-the-counter medication (Azo-Gesic, Baridium, Urinary Pain Relief) that has been used safely for decades as a bladder analgesic and taints the urine orange.

Over the past few months, increasing evidence suggests that phenazopyridine may reduce transient postoperative urinary retention. Transient urinary retention is common after urogynecologic surgery and is assessed postoperatively by performing a void trial (VT) prior to discharge. In a study designed to determine the time from administration of oral phenazopyridine to visualize dye from the ureters, Propst et al incidentally found that 38% of patients (19 of 49) failed postoperative VTs without phenazopyridine, but only 19% (9 of 47) failed with phenazopyridine, p=0.04. Most recently, a study by Duenas-Garcia et al designed to examine local anesthetics and urinary retention in subjects undergoing midurethral slings found that phenazopyridine decreased the VT failure rate from 30% to 8% (5). The investigators hypothesize that giving a dose of phenazopyridine the morning after surgery will significantly reduce the rate of postoperative urinary retention in women undergoing prolapse repair.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing overnight admission after prolapse surgery

Exclusion Criteria:

* Unable to provide consent
* Under 18 years of age
* Pregnant women
* Prisoners
* Using intermittent self-catheterization preoperatively
* Neurological disease or spinal cord injury resulting in voiding dysfunction
* Undergoing spinal or epidural anesthesia for the procedure
* Allergy to phenazopyridine
* Renal insufficiency
* Liver disease
* Intra-operative bladder injury necessitating use of prolonged indwelling Foley catheter

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Flynn, MD, Principal Investigator — UMass Worcester
Locations (1):
- University of Massachusetts, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sierra T, Taylor DL, Leung K, Hall CD, Flynn MK. The Effect of Phenazopyridine on Immediate Postoperative Voiding After Prolapse Surgery: A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):85-89. doi: 10.1097/SPV.0000000000000737. PMID 31033527

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenazopyridine on POD1: Participant is given Phenazopyridine 200 mg on postoperative day 1
  76 subjects were randomized into this arm
  4 were removed from the intent-to-treat analysis:
  * 1 had a bowel injury re-operation that precluded performing a void trial
  * 1 intraoperative cystotomy that precluded performing a void trial
  * 2 were using Foley catheters preoperatively, which was part of the exclusion criteria
    72 subjects in the intent-to-treat analysis
    3 did not receive the intervention:
  * 1 was too nauseous
  * 1 was erroneously missed
  * 1 refused
    69 subjects in the as-treated analysis
- No Intervention on POD1: Subject is not given Phenazopyridine on postoperative day 1
  76 subjects were randomized into this arm
  2 were removed from the intent-to-treat analysis:
  * 1 intraoperative cystotomy that precluded performing a void trial
  * 1 had spinal anesthesia, which was part of the exclusion criteria
    74 subjects in the intent-to-treat analysis
    3 cross-overs were brought in from the intervention arm because they did not receive the medication
    77 subjects in the as-treated analysis
Period: Overall Study
Arm/Group | Phenazopyridine on POD1 | No Intervention on POD1
Started | 76 | 76
Intent-to-treat Analysis | 72 | 74
As-treated Analysis | 69 | 77
Completed | 76 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phenazopyridine: Participant is given Phenazopyridine on morning of postoperative day 1
- No Phenazopyridine: Participant is not given Phenazopyridine on morning of postoperative day 1
- Total: Total of all reporting groups
Arm/Group | Phenazopyridine | No Phenazopyridine | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (12.8) | 60.9 (13.5) | 61.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 76 | 152
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61 | 59 | 120
  Non-white | 14 | 17 | 31
  Declined to answer | 1 | 0 | 1
Concomitant hysterectomy [Count of Participants; unit: Participants] | 59 | 62 | 121

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Urinary Retention After Pelvic Organ Prolapse Surgery (INTENT-TO-TREAT)
Description: Rate of postoperative urinary retention after pelvic organ prolapse surgery as determined by those who failed a standardized void trial. A successful void trial is defined as a postvoid residual of less than half of the voided volume.
Time Frame: postoperative day 1
Population: Intent-to-treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Phenazopyridine | No Phenazopyridine
Number analyzed (Participants) | 72 | 74
Participants | 30 | 25

2. Other Pre Specified Outcome: Number of Participants With Postoperative Urinary Retention After Pelvic Organ Prolapse Surgery (AS-TREATED)
Description: as for outcome 1
Time Frame: postoperative day 1
Population: As-treated analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Phenazopyridine | No Phenazopyridine
Number analyzed (Participants) | 69 | 77
Participants | 28 | 27

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Phenazopyridine: Participant is given Phenazopyridine
  Phenazopyridine: Phenazopyridine on morning of postoperative day 1
  76 subjects were randomized into this arm
  4 were removed from the intent-to-treat analysis:
  * 1 had a bowel injury re-operation that precluded performing a void trial
  * 1 intraoperative cystotomy that precluded performing a void trial
  * 2 were using Foley catheters preoperatively, which was part of the exclusion criteria
    72 subjects in the intent-to-treat analysis
    3 did not receive the intervention:
  * 1 was too nauseous
  * 1 was erroneously missed
  * 1 refused
    69 subjects in the as-treated analysis
- No Phenazopyridine: Participant is not given Phenazopyridine
  76 subjects were randomized into this arm
  2 were removed from the intent-to-treat analysis:
  * 1 intraoperative cystotomy that precluded performing a void trial
  * 1 had spinal anesthesia, which was part of the exclusion criteria
    74 subjects in the intent-to-treat analysis
    3 cross-overs were brought in from the intervention arm because they did not receive the medication
    77 subjects in the as-treated analysis
Arm/Group | Phenazopyridine | No Phenazopyridine
All-Cause Mortality (participants affected / at risk) | 1/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/76 | 0/76
Other Adverse Events (participants affected / at risk) | 9/76 | 14/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenazopyridine (N=76) | No Phenazopyridine (N=76)
Bowel injury re-operation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Re-operation and ICU admission for bowel injury during prolapse surgery
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenazopyridine (N=76) | No Phenazopyridine (N=76)
Urinary tract infection (Infections and infestations) | 9 (9) | 14 (14) — A positive urine culture, urinalysis, or antibiotic treatment within 6 weeks postoperatively constituted a UTI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03065075/Prot_SAP_000.pdf